CLINICAL TRIAL: NCT07147998
Title: Assessing the Impact of 2D:4D Ratio on Oral Hygiene Performance and Gingival Health
Brief Title: Impact of 2D:4D Ratio on Oral Hygiene and Gingival Health
Status: Completed | Type: Observational
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Ekin Besiroglu, Assist. Prof., Okan University
Other Study IDs: 2023/165-01
Record Dates: First submitted 2025-08-08; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Oral Hygiene; Gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Oral hygiene instruction — Oral hygiene and gingival health of all patients were assessed using the Turesky Modification of the Quigley-Hein Plaque Index and the Gingival Index. Tooth brushing frequency was recorded. The 2D:4D ratio was calculated by dividing the second digit length by the fourth, with three measurements taken per finger to ensure reliability. A cut-off value of 1 was used to evaluate prenatal androgen influence, and participants were grouped by 2D:4D ratio (≥1 or <1). All participants received standardized oral hygiene instructions from the same instructor, including Modified Bass brushing and interdental cleaning. A second clinical exam was performed one week later by the same examiner, and both indices were re-scored.

SUMMARY:
The second-to-fourth digit ratio (2D:4D)-the ratio of the length of the index finger to that of the ring finger-has gained increasing attention as a non-invasive, stable biomarker of prenatal sex hormone exposure. The 2D:4D ratio is believed to reflect the balance of prenatal androgens (especially testosterone) and estrogens. Lower ratios (more masculinized) indicate higher prenatal testosterone exposure, whereas higher ratios (more feminized) are associated with lower testosterone and higher estrogen levels. Research has linked variations in 2D:4D to a broad spectrum of behavioral traits, cognitive abilities, and health outcomes. 2D:4D has been shown to have strong associations with motor performance, especially skills that require fine motor coordination. However, while many studies have examined the role of 2D:4D in sports and cognition, its relationship to health-related behaviors involving motor skills remains underexplored. One such domain is oral hygiene, which requires sustained fine motor coordination-particularly in actions like tooth brushing and flossing. Despite the clear motor demands of such behaviors, the potential connection between 2D:4D and oral hygiene has not yet been systematically investigated. This study aims to fill this gap by exploring the association between the 2D:4D digit ratio and oral hygiene practices.

DETAILED DESCRIPTION:
Background and Rationale The second-to-fourth digit ratio (2D:4D)-the ratio of the length of the index finger to that of the ring finger-is a morphological index thought to reflect prenatal sex-hormone exposure. The trait is determined during early fetal development and is generally stable from early childhood into adulthood. Prior research has examined associations between 2D:4D and behavioral, cognitive, and motor outcomes in various populations; however, the relationship between 2D:4D and everyday health behaviors that require fine motor coordination (e.g., tooth brushing and interdental cleaning) has not been comprehensively evaluated. This study is designed to test whether 2D:4D is associated with oral hygiene measures and practices.

Objectives and Hypotheses Primary objective: To evaluate the association between right-hand 2D:4D and dental plaque accumulation as measured by the Turesky Modification of the Quigley-Hein Plaque Index (QHPI) and the Löe-Silness Gingival Index (GI) at baseline and after standardized oral-hygiene instruction.

Secondary objectives: (1) To examine whether sex and hand dominance modify the association between 2D:4D and oral-hygiene outcomes; (3) To explore whether baseline 2D:4D is related to self-reported brushing frequency.

Hypotheses (a priori): Lower 2D:4D (putatively reflecting higher prenatal androgen exposure) will be associated with differences in oral-hygiene performance compared with higher 2D:4D. Direction and magnitude will be tested empirically.

Study Design and Setting This is a single-center, observational study with a baseline assessment and a planned follow-up visit approximately 7 days after standardized instruction. The study will be conducted in the Periodontology Clinic of the Faculty of Dentistry at Istanbul Okan University.

Participants Adults aged 18-56 years who attend the clinic for routine examination and provide written informed consent will be eligible. Key exclusion criteria will include conditions that could interfere with hand measurements or oral-hygiene procedures (e.g., hand injuries affecting the right index or ring finger, severe periodontal disease requiring urgent treatment, or systemic conditions judged by investigators to preclude participation). The planned sample size is approximately 126 participants, based on an a priori power calculation (two-tailed; α = 0.05; power [1 - β] = 0.80).

Procedures At the initial visit (Day 0), socio-demographic data will be recorded. Oral hygiene and gingival status will be assessed using the QHPI and GI, respectively. Brushing frequency will be recorded by self-report. All teeth except third molars will be scored on buccal and lingual surfaces. Dental plaque will be disclosed with Mira-2-Ton Disclosing Solution (Hager & Werken, Germany) prior to QHPI scoring.

The lengths of the second (index) and fourth (ring) digits on the right hand will be measured on the ventral surface using a digital caliper, from the fingertip to the midpoint of the basal crease. Three measurements will be taken for each finger and averaged; the 2D:4D ratio will be computed as (2D length)/(4D length). For exploratory analyses, a prespecified cut-off of 1.0 will be used to define subgroups (2D:4D < 1.0 vs ≥ 1.0) within each sex.

Following baseline assessments, all participants will receive standardized oral-hygiene instruction from the same instructor, including the Modified Bass brushing technique and the use of dental floss or interdental brushes. A follow-up visit will occur approximately 7 days later (Day 7 ± 2), at which QHPI and GI will be reassessed by the same examiner.

Quality Control To minimize inter-examiner variability, all digit and oral-hygiene measurements will be performed by a single examiner who will undergo standardized training and calibration before data collection. Calibration will continue until predefined reproducibility thresholds for both measurement types are met.

Outcome Measures Primary outcome: QHPI score (0-5) per tooth surface, aggregated per participant at Day 0 and Day 7.

Secondary outcomes: GI score (0-3) per site, aggregated per participant at Day 0 and Day 7; self-reported brushing frequency (times/day).

Statistical Analysis Plan Descriptive statistics will be presented as Mean ± Standard Error (SE) or appropriate alternatives. Assumptions for parametric testing will be evaluated using the Shapiro-Wilk test (normality) and Levene's test (homogeneity of variance). Between-group comparisons of 2D:4D by sex and hand dominance will use Student's t-tests when assumptions are met.

To assess changes over time and the effects of prespecified factors (sex, hand dominance, and 2D:4D subgroup), two-way mixed-design ANOVA models (time: Day 0 vs Day 7; between-subject factors as specified) will be applied to QHPI and GI. When significant main effects or interactions are observed, pairwise comparisons will use a Bonferroni adjustment. Pearson correlation will be used to examine associations between continuous 2D:4D and oral-hygiene measures. All tests will be two-sided with α = 0.05. Analyses will be performed using SPSS version 30 or later.

Ethics The protocol will be conducted in accordance with the Declaration of Helsinki and has received approval from the relevant institutional ethics committee. Written informed consent will be obtained from all participants before enrollment.

ELIGIBILITY:
Inclusion Criteria:

Systemically healthy University graduates or currently enrolled in a university program Presence of 28 natural teeth No orthodontic appliances or crown restorations in the oral cavity Non-smokers No previous oral hygiene instruction from a dental professional Clinical diagnosis of gingivitis

Exclusion Criteria:

Presence of any systemic disease or condition that may affect periodontal health Not a university graduate and not currently enrolled in a university program Fewer than 28 natural teeth Orthodontic appliances or crown restorations present in the oral cavity Current smokers Previous oral hygiene instruction from a dental professional Clinical diagnosis of periodontitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults over 18 years of age, systemically healthy, without psychological or neurological disorders, able to cooperate during examinations and procedures, university students or graduates, with at least 28 natural teeth, non-smokers, with no fixed orthodontic appliances or crown prostheses, no prior oral hygiene education from a dental professional, and a clinical diagnosis of gingivitis.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Mean Quigley-Hein Plaque Index Score (Turesky Modification) | Baseline (Day 0) and 1 week after oral hygiene instruction.
  Dental plaque will be scored on buccal and lingual surfaces of all teeth except third molars using the Turesky Modification of the Quigley-Hein Plaque Index (scale 0-5; 0 = no plaque, 5 = plaque covering ≥ two-thirds of crown). Scores per tooth will be averaged per participant.
Mean Löe-Silness Gingival Index Score | Baseline (Day 0) and 1 week after oral hygiene instruction.
  Gingival inflammation will be assessed on buccal and lingual surfaces at mesial, mid-buccal, and distal sites using the Löe-Silness Gingival Index (scale 0-3; 0 = healthy, 3 = severe inflammation with spontaneous bleeding). Scores will be averaged per participant.

SECONDARY OUTCOMES:
Right-hand 2D:4D Digit Ratio | Baseline (Day 0)
  Lengths of the index (2D) and ring (4D) fingers of the right hand will be measured three times using a digital caliper (ventral surface, fingertip to basal crease). The mean lengths will be used to calculate the 2D:4D ratio.
Self-reported Tooth Brushing Frequency | Baseline (Day 0)
  Participants will report their average number of daily tooth brushing episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Ekin Beşiroğlu Turgut, Study Director — Okan University
Locations (1):
- İstanbul Okan University, Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided